CLINICAL TRIAL: NCT02589691
Title: Addition of Neuromuscular-Blocking Agents During Sevoflurane Induction in Infants : Potential Interest in Reducing Hypoxemia Episodes
Brief Title: Neuromuscular-Blocking Agents and Hypoxemia During Intubation in Infants (ROC-HYPOX)
Acronym: ROC-HYPOX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FDE_2014_25
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-03

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia | interventions — Rocuronium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rocuronium (Experimental): Intra-venous injection during induction anesthesia of 0.3 mg/kg (1 mL/kg) of rocuronium
  Interventions: Drug: Rocuronium
- Placebo (Placebo Comparator): Intra-venous injection during induction anesthesia of 1 mL/kg of sodium chloride 0.9%
  Interventions: Other: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Rocuronium
  Arms: Rocuronium
Other: Sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
The prevention of the occurrence of respiratory events is a constant concern in pediatric anesthesia, as these represent the main cause of the anesthesic mortality. These events occur partly during induction of anesthesia and are all the more frequent as the child is young.

The French recommendations do not propose the use of neuromuscular-blocking agents in pediatric anesthesia. This recommendation is controversial In a recently published study, it has been shown that the use of neuromuscular blocking agents during induction in children under 2 years improves intubating conditions and reduces the incidence of hemodynamic and respiratory events. This monocentric study, centered on intubating conditions, does not allow to conclude on the influence of muscle relaxants on reduction of the respiratory morbidity.

The objective of study is to demonstrate that, in children under 2 years, changing the anesthesia protocol can reduce the incidence and severity of episodes of hypoxemia associated with respiratory events occurring during induction

ELIGIBILITY:
Inclusion Criteria:

* age <2 years
* indication of general anesthesia with tracheal intubation
* inhalational induction scheduled
* written informed consent of both parents

Exclusion Criteria:

* contra-indication to inhalational induction (full stomach)
* contra-indication to the use of rocuronium
* American Society of Anesthesiologists score (ASA) III or IV
* intracranial surgery
* parental refusal
* absence of affiliation to social security

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 412 (Estimated)
Dates: Start 2015-12-23 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence, expressed as a percentage, of at least on episode of hypoxemia, defined as an arterial oxygen saturation <90%, obtained by continuous measurement of pulse oximetry. | Up to 15 minutes after anesthesia induction

SECONDARY OUTCOMES:
Cumulative duration of hypoxemia expressed in seconds and defined as an arterial oxygen saturation <90% | Up to 15 minutes after anesthesia induction
Cumulative duration, expressed in seconds, with a decreased in arterial oxygen saturation of 5% as compared to the arterial oxygen saturation at baseline | Up to 15 minutes after anesthesia induction
Lowest recorded value of arterial oxygen saturation. | Up to 15 minutes after anesthesia induction
Incidence, expressed as a percentage, of at least one episode of bronchospasm | Up to 15 minutes after anesthesia induction
Incidence, expressed as a percentage, of at least one episode of laryngospasm | Up to 15 minutes after anesthesia induction
Duration, expressed in seconds, of apnea | Up to 15 minutes after anesthesia induction

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Hospitalier Intercommunal Creteil (CHIC), Créteil
  - Hôpital Jeanne de Flandre, CHRU de Lille, Lille
  - Hôpital Necker-Enfants malades, Paris
  - Hopital Robert Debre, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - CHU de Toulouse, Toulouse